CLINICAL TRIAL: NCT03263156
Title: Effects of a Brief Parent-based Sleep Intervention for Children With Attention Deficit Hyperactivity Disorder
Brief Title: A Brief Parent-based Sleep Intervention for ADHD Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Shirley Xin Li, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30160604
Record Dates: First submitted 2017-08-23; First posted 2017-08-28 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: ADHD; Insomnia
Keywords: sleep; ADHD; behavioural intervention; insomnia
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention will involve two face-to-face consultation sessions and one follow-up phone call with parents to help them learn sleep hygiene practices and specific behavioural strategies to improve their child's sleep and follow up on the progress.
  Interventions: Behavioral: Sleep hygiene practices and behavioural intervention
- Waiting-list control (No Intervention): Children in the waiting-list control group will receive usual clinical care.

INTERVENTIONS:
Behavioral: Sleep hygiene practices and behavioural intervention — The first session will involve the provision of sleep-related psycho-education (e.g. sleep hygiene practices) and specific strategies to tackle problematic sleep-related behaviours, as well as collaborative goal setting and development of management plan tailored to the child's sleep problem for the next two weeks. The second session will involve a review of the sleep diary and a reinforcement of learned strategies, and focus on problem-solving to tackle any issues that have emerged from implementing the behavioural strategies at home. A follow-up phone call will be made two weeks later to provide parents with an opportunity to ask any further questions and to consolidate learned strategies and further troubleshoot.
  Arms: Intervention group

SUMMARY:
Sleep problems are very common in children with ADHD, with a prevalence rate as high as 73%, and often pose significant challenges and stress to the families. Sleep problems in ADHD children are strongly associated with the exacerbation of daytime symptoms, impaired physical health, and poor parental mental health. The present study is a randomised controlled trial to compare the effects of a parent-based sleep intervention for children with ADHD (aged 6-12). Eligible participants will be randomised to either intervention (two face-to-face consultation sessions and one follow-up phone call) or waiting-list control condition. Assessments will be conducted at pre-treatment (baseline), one-week after the intervention (post-treatment), and 3 months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6-12 years old;
* With a clinical diagnosis of ADHD (any subtype), as confirmed by the Diagnostic Interview Schedule for Children-version-IV (DISC-IV);
* With parent-reported insomnia (difficulty initiating sleep and/or maintaining sleep).

Exclusion Criteria:

* Children with a serious medical condition (e.g. severe cerebral palsy) or intellectual disability (IQ<70);
* Children with a neurological and/or medical condition that may lead to disordered sleep;
* Suspected clinical sleep disorders (e.g. obstructive sleep apnea, OSA) that may potentially contribute to a disruption in sleep continuity and quality, as assessed by the Children's Sleep Habits Questionnaire (CSHQ). If the child is suspected of a clinical sleep disorder, he/she will be referred to appropriate services;
* Children who are already receiving specialised help (behavioural intervention) for their sleep from a psychologist or at a specialized sleep clinic.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Child: Change of child's sleep | Baseline, 1-week and 3-month posttreatment
  Change of the child's sleep measured by the Children's Sleep Habits Questionnaire (CSHQ), and sleep problems rated by parent (none, mild, moderate, severe)

SECONDARY OUTCOMES:
Child: Change of daytime sleepiness | Baseline, 1-week and 3-month posttreatment
  Pediatric Daytime Sleepiness Scale (PDSS) - parent report
Child: Change of other sleep measures | Baseline, 1-week and 3-month posttreatment
  Daily sleep diary and actigraphic assessment for consecutive seven days
Child: Change of ADHD symptoms | Baseline, 1-week and 3-month posttreatment
  Strengths and Weaknesses of ADHD Symptoms (SWAN) - parent report
Child: Change of child's behaviour & other clinical symptoms | Baseline, 1-week and 3-month posttreatment
  Strengths and Difficulties Questionnaire - parent report; Child Behavior Checklist (CBCL) - parent report
Child: Change of quality of life | Baseline, 1-week and 3-month posttreatment
  Pediatric Quality of Life Inventory 4.0 - parent proxy report (PedsQL) - parent report
Child: Change of cognitive performance (sustained attention) | Baseline, 1-week and 3-month posttreatment
  Continuous Performance Test (CPT)
Child: Change of cognitive performance (auditory attention span) | Baseline, 1-week and 3-month posttreatment
  Digit Span
Child: Change of cognitive performance (working memory) | Baseline, 1-week and 3-month posttreatment
  N-back
Child: Change of cognitive performance (cognitive processing) | Baseline, 1-week and 3-month posttreatment
  Letter-digit substitution task
Child: Change of cognitive performance (cognitive flexibility) | Baseline, 1-week and 3-month posttreatment
  Bergs Card Sorting Test (BCST)
Child: Change of cognitive performance (planning skills) | Baseline, 1-week and 3-month posttreatment
  Tower of London (TOL)
Change of parental self-reported sleep quality | Baseline, 1-week and 3-month posttreatment
  Pittsburgh Sleep Quality Index (PSQI)
Change of parental insomnia symptoms | Baseline, 1-week and 3-month posttreatment
  Insomnia Severity Index (ISI)
Change of parental daytime sleepiness | Baseline, 1-week and 3-month posttreatment
  Epworth Sleepiness Questionnaire (ESS)
Change of parental sleep parameters as measured by actigraphy | Baseline, 1-week and 3-month posttreatment
  Actigraphic sleep parameters
Change of parental sleep hygiene practice | Baseline, 1-week and 3-month posttreatment
  Sleep Hygiene Index (SHI)
Change of parental stress | Baseline, 1-week and 3-month posttreatment
  Parental Stress Index - Short Form (PSI-SF)
Change of parental mood symptoms | Baseline, 1-week and 3-month posttreatment
  Depression Anxiety Stress Scales - 21 item (DASS-21)
Change of parental daytime fatigue | Baseline, 1-week and 3-month posttreatment
  Multidimensional Fatigue Inventory (MFI)
Parent's satisfaction to the treatment | Baseline, 1-week and 3-month posttreatment
  Treatment satisfaction rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Xin Li, PhD,DClinPsy, Principal Investigator — Department of Psychology, The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Child and Adolescent Psychiatric Service Clinic, New Territories East Cluster (NTEC), Hospital Authority, Hong Kong
  - Sleep Research Clinic & Laboratory, Department of Psychology, The University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2016-09-29): https://cdn.clinicaltrials.gov/large-docs/56/NCT03263156/Prot_001.pdf